CLINICAL TRIAL: NCT05438017
Title: Assessment of the Performance of the Dreem 3 System for EEG Sleep Monitoring in the Lab Setting
Brief Title: Performance Evaluation of the Dreem 3 System for Sleep Assessment in Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dreem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OCTAVE 3
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Insomnia
Keywords: Dreem; Insomnia symptoms; Sleep; Polysomnography; Performance; EEG; Sleep monitoring
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Dreem + PSG (Experimental)
  Interventions: Device: Dreem 3 System vs PSG

INTERVENTIONS:
Device: Dreem 3 System vs PSG — Dreem 3 System to be worn by each participant while undergoing in-lab sleep study with PSG.

SUMMARY:
The objective of the clinical investigation is to assess the performance of the Dreem 3 System for sleep assessment compared to a FDA-cleared PSG assessment and human sleep expert scoring in a population experiencing insomnia symptoms.

DETAILED DESCRIPTION:
Subjects enrolled in the study will come to the sleep laboratory around 8 pm. Their involvement in the protocol will only require them to be equipped by the technician with Dreem 3 in addition to the PSG reference system. This involves the technician placing all the PSG electrodes on the subject's head as per normal practice, and then positioning the Dreem 3 headband so that both devices can operate simultaneously. The subject will be allowed to go to his/her room and do quiet activities (reading, film watching, chatting) prior to sleeping. At the end of the night, the technician will remove the Dreem 3 headband and the PSG.

A technical quality control will be performed on the collected data in accordance with the standard operating procedures, as defined in the study protocol. Recordings that do not meet the quality control criteria will be excluded from further analysis.

Subjects will receive the PSG report at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 22 and ≤ 70 years old inclusive.
* Able to read, understand and sign an informed consent form.
* Subjects with stable disease or/and taking stable medications for at least 2 months can be included under Principal Investigator or Sub-Investigator discretion
* Self-reported insomnia symptoms (by means of a questionnaire completed by the participant before their visit to the sleep lab) as defined by International Classification of Sleep Disorders, third edition (ICSD-3), confirmed by a clinician.

Exclusion Criteria:

* Female subjects who are pregnant, or breastfeeding.
* Subject under 22 and above 70 years old inclusive.
* Not able to read, understand and sign an informed consent form
* Subjects with BMI ≥ 40
* Taking medications that induce somnolence or wakefulness, or that can interfere with sleep recording:

  * If the subject is taking OTC medications that can induce somnolence or wakefulness, he/she must not take it the day of the measurement.
  * Prescription only drugs that induce somnolence or wakefulness must be stopped one week before, as PI or Sub-I discretion and/or review with subject's physician.
* Subjects previously diagnosed with Obstructive Sleep Apnea (OSA), REM Sleep Disorder, Narcolepsy, Hypersomnia, or significant difficulty breathing due to underlying condition(s), or subjects diagnosed with Central Nervous System (CNS) disease.
* Subjects that suffer from an unstable disease
* Any incidental finding on the Polysomnography reference system, happening during the study recording, that interferes with eligibility (probable moderate/severe undiagnosed OSA)
* Subjects who may experience fitting difficulties with the headband, including people with head circumference < 53cm, or a hairstyle impeding the sensor placement (tight braids, hair extension, dreadlocks…) as determined by the investigator.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Performance of the automatic sleep stage scoring of the Dreem 3 System compared to the consensus of 3 independent certified sleep scorers realized on the polysomnography signal. | Day 1

SECONDARY OUTCOMES:
TST (Total Sleep Time) | Day 1
  Total time (in minutes) the subject spends asleep (TST) as automatically determined by the Dreem 3 System compared to the TST determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
SE (Sleep Efficiency) | Day 1
  Sleep efficiency (%) as automatically determined by the Dreem 3 System compared to the sleep efficiency determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
SOL (Sleep Onset Latency) | Day 1
  Sleep Onset Latency (in minutes) as automatically determined by the Dreem 3 System compared to the sleep onset latency determined by the consensus of 3 certified sleep scorers's scoring of the subject's PSG record from the same night.
LPS (Latency to Persistent Sleep) | Day 1
  Latency to Persistent Sleep (in minutes) as automatically determined by the Dreem 3 System compared to the latency to persistent sleep determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
WASO (Wake After Sleep Onset) | Day 1
  Total time (in minutes) the subject spends awake from sleep onset to final epoch of sleep (WASO) as automatically determined by the Dreem 3 System compared to the WASO determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
Total time spent in N2 sleep stage | Day 1
  Total time (in minutes) the subject spends in AASM N2 sleep stage as automatically determined by the Dreem 3 System compared to the N2 time determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
Total time spent in N3 sleep stage | Day 1
  Total time (in minutes) the subject spends in AASM N3 sleep stage as automatically determined by the Dreem 3 System compared to the N3 time determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
Total time spent in REM sleep stage | Day 1
  Total time (in minutes) the subject spends in AASM REM sleep stage as automatically determined by the Dreem 3 System compared to the REM time determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
Total time spent in N1 sleep stage | Day 1
  Total time (in minutes) the subject spends in AASM N1 sleep stage as automatically determined by the Dreem 3 System compared to the N1 time determined by the consensus of 3 certified sleep scorers' scoring of the subject's PSG record from the same night.
Respiratory Rate | Day 1
  Respiratory rate for each 30 second epoch (in cycles per minute) computed by the accelerometer of the Dreem device compared to the respiratory rate computed by the PSG sensor.

CONTACTS AND LOCATIONS:
Locations (2):
- Biotrial Inc, Newark, New Jersey, United States
- Biotrial Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No